CLINICAL TRIAL: NCT02150135
Title: Effect of Oncothermia on Improvement of Quality of Life in Unresectable Pancreatic Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hospicare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jin-Hyeok Hwang, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-IMGPB-2014-02
Record Dates: First submitted 2014-05-24; First posted 2014-05-29 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Cancer, Pancreas
Keywords: Pancreatic cancer; Quality of life; Pain
MeSH Terms: conditions — Pancreatic Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oncothermia group (Experimental): Patients were treated with oncothermia 2 or 3 times a week. Treatment was performed for about 1 hours per each visits.
  Interventions: Other: Oncothermia

INTERVENTIONS:
Other: Oncothermia — Oncothermia is a kind of hyperthermia treatment. It serves heat energy more selectively than conventional hyperthermia.

SUMMARY:
Patients with pancreatic cancer often suffer from pain. Because of such a pain, their quality of life have seriously deteriorated. There have been a few studies that showed an effect for pain control by hyperthermia (heating the patient's body). However, there are several limitations in conventional hyperthermia. In this study, the investigators tried to show the effect of "Oncothermia" which is more selective to malignant tissue than conventional hyperthermia for pain control, increasing quality of life, and anti-tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable or recurred pancreatic ductal adenocarcinoma
* After the each cycle of chemotherapy, the disease status was "stable disease"

Exclusion Criteria:

* Person who has an experience of hyperthermia treatment
* Person who has a difficulty of sensing heat
* Person who has a skin graft or breast reconstruction surgery
* Person who has a cardiac pacemaker or an implanted metal
* Pregnant or breast feeding women
* Person with uncontrolled infection, diabetes, hypertension, ischemic heart disease, myocardial infarct within 6 months
* Person who was treated with unproved drugs within 6 months
* Person who have a serious disease which can affect the person's safety
* Person who do not consent to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
ECOG score change | 3 months after oncothermia treatment

SECONDARY OUTCOMES:
Progression free survival rate | 3 months later after oncothermia treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hyeok Hwang, MD PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea